CLINICAL TRIAL: NCT06142838
Title: Community Pharmacist Intervention to Enhance Adherence in Cardiovascular Drug Initiators
Acronym: PHARM-ADHERE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Vrije Universiteit Brussel (Other); Université de Liège (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B6702023000469 - ONZ-2023-0360
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; Cardiovascular Disease Prevention
Keywords: Medication adherence
MeSH Terms: conditions — Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Community pharmacist intervention
  Interventions: Behavioral: community pharmacist intervention
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Behavioral: community pharmacist intervention — The community pharmacist intervention comprises 2 parts: (1) first prescription counseling (oral and written information), and (2) a follow-up consultation (by telephone or in person) 7-14 days later, to identify problems with adherence/treatment
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to evaluate a community pharmacist intervention aimed at improving medication adherence in patients starting newly prescribed medication for cardiovascular disease prevention. The main questions it aims to answer are:

* Does this community pharmacist intervention improve medication adherence?
* Which patients benefit the most from the intervention?
* How do patients experience the start-up of newly prescribed medication (which questions do they have and do they experience side effects?)?
* How do patients and pharmacists experience the intervention?

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a first prescription for one of the following drug classes: antihypertensive drugs (= low-ceiling diuretics, beta blocking agents (excl. non-selective beta-blocking agents), ACE inhibitors, angiotensin II receptor blockers, calcium channel blockers), lipid-lowering drugs (= statins), antidiabetic drugs (= metformin, glucagon-like peptide-1 (GLP-1) analogues, sodium-glucose co-transporter 2 (SGLT2) inhibitors), or any combination thereof.
* Age 18 years or older
* Community-dwelling

Exclusion Criteria:

* The drug is prescribed for a non-cardiovascular indication (e.g. beta-blocking agent for migraine prophylaxis)
* Communication with the patient is not possible (e.g. due to cognitive impairment, insufficient knowledge of Dutch or French language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
NIH Patient Reported Outcomes Measurement Information System (PROMIS) Medication Adherence Scale (PMAS) | At 6 weeks and at 12 weeks follow-up
  Patient-reported measure of medication adherence

SECONDARY OUTCOMES:
Medication Possession Ratio (MPR) | Over 26 weeks post-baseline
  Measure of medication adherence, using pharmacy refill records
Discontinuation rate | Over 26 weeks post-baseline
  % of patients discontinuing the medication
Medication knowledge questionnaire | At 6 weeks and at 12 weeks follow-up
  Questionnaire evaluating patient's basic knowledge about the medication
Beliefs about Medicines Questionnaire (BMQ-Specific) | At 6 weeks and at 12 weeks follow-up
  Questionnaire evaluating patient's beliefs about the necessity of prescribed medication for controlling their illness (Specific-Necessity) and their concerns about the potential adverse consequences of taking it (Specific-Concerns)
Treatment response | At baseline and at 12 weeks follow-up
  Systolic and diastolic blood pressure for patients starting an antihypertensive drug; lipid levels (total cholesterol, LDL and HDL) for patients starting a lipid-lowering drug; HbA1c for patients starting an antidiabetic drug
Healthcare utilization | Over 12 weeks post-baseline
  Number of general practitioner (GP) visits, specialist-physician visits, emergency department (ED) visits and hospital admissions

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Care Unit (Ghent University), Ghent, Belgium